CLINICAL TRIAL: NCT04431414
Title: A Prospective Study of Acute Immune Responses to SARSCoV-2 Infection
Brief Title: A Study of Immune Responses to the Virus That Causes COVID-19
Acronym: CoVPN 5001
Status: Completed | Type: Observational
Sponsor: COVID-19 Prevention Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CoVPN 5001; 5UM1AI068614-14 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Persons that are positive for SARS-CoV-2 and are asymptomatic
  Interventions: Other: Sample collection
- Group 2: Persons that are positive for SARS-CoV-2 with recent onset of mild symptoms (not hospitalized)
  Interventions: Other: Sample collection
- Group 3: Persons that are positive for SARS-CoV-2 and are symptomatic hospitalized patients
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — * blood, nasal swab, nasal wash, and saliva
  * optional stool swab

SUMMARY:
The purpose of this study is to learn more about the acute response to infection with and recovery from the virus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Some people know this virus by the name "coronavirus." It can cause the disease called COVID-19.

The information gained from the study can be used to help develop better tests for SARS-CoV-2 infection and COVID-19 disease and may help in developing future vaccines, other prevention strategies, and treatments.

DETAILED DESCRIPTION:
This is a prospective study of acute immune responses to SARSCoV-2 infection.

The study will include 3 groups, as described in the table below. Groups are defined based on clinical status at enrollment, but for the purposes of data analysis, participants who experience disease progression can contribute data to other cohorts.

Participants will complete six visits over 28 days followed by a health contact at Month 2 (one month after the last scheduled visit). Additional follow up visit(s) may be added over time in response to evolving information regarding SARS-CoV-2 infection and COVID-19.

Study visits may include review of medical history; interviews/questionnaires; pregnancy tests (for participants assigned female sex at birth); blood draws; nasal swab, nasal wash, and saliva sample collection; and optional stool sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Test result indicating presence of SARS-CoV-2 virus. Sites must have results from assays that are approved as FDA-emergency use authorized or as standard-of-care by other applicable regional governing bodies. For timing of testing, please see group specific criteria below.
* Ability and willingness to provide informed consent.
* Willingness to have clinical research staff come to place of residence or hospital if needed.
* Willingness to be followed for the planned duration of the study.
* Assessment of understanding: volunteer demonstrates understanding of this study.
* Agreement to allow access to medical records.
* Asymptomatic participants:

  * No current symptoms.
  * No symptoms consistent with COVID-19 within 2 weeks prior to positive test according to the clinical judgement of the investigating clinician. Symptoms include, but are not limited to, fever, headache, sore throat, cough, dyspnea, rhinorrhea, diarrhea, myalgias, chills, and anosmia. Please refer to https://www.cdc.gov/coronavirus/2019-ncov/symptomstesting/symptoms.html for the current list of symptoms consistent with COVID-19.
  * Positive SARS-CoV-2 RNA test or antigen test within six days prior to enrollment (target time) up to 10 days prior to enrollment (upper allowable window).
* Symptomatic (non-hospitalized) participants:

  * Onset of mild symptoms consistent with COVID-19 within 6 days prior to enrollment (target time) up to 14 days prior to enrollment (upper allowable window). Symptoms of COVID-19 to be determined by the clinical judgement of the investigating clinician including-- but not limited to-- fever, headache, sore throat, cough, dyspnea, rhinorrhea, diarrhea myalgias, chills, and anosmia. Please refer to https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html for the current list of symptoms consistent with COVID-19.
  * Positive SARS-CoV-2 RNA test or antigen test within six days prior to enrollment (target time) up to 10 days prior to enrollment (upper allowable window).
* Symptomatic (hospitalized) participants

  * Participant hospitalized for COVID-19 within 3 days prior to enrollment (note: there is no timeframe for either symptom onset or timing of SARS-CoV-2 PCR or antigen testing for hospitalized participants)

Exclusion Criteria:

* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or a volunteer's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have tested positive for SARSCoV-2 virus by RT-PCR or antigen testing.
Sampling Method: Probability Sample
Enrollment: 953 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Response rate of SARS-CoV-2-specific B cells in peripheral blood samples | Measured through day 14
  Characterized using fluorescently labeled recombinant proteins in combination with a flow cytometry phenotyping panel
Magnitude of SARS-CoV-2-specific B cells in peripheral blood samples | Measured through day 14
  Characterized using fluorescently labeled recombinant proteins in combination with a flow cytometry phenotyping panel
Phenotypic characterization of SARS-CoV-2-specific B cells in peripheral blood samples | Measured through day 14
  Characterized using fluorescently labeled recombinant proteins in combination with a flow cytometry phenotyping panel
Response rate of SARS-CoV-2-specific antibody binding in serum samples | Measured through day 28
  Measured by binding antibody multiplex assay (BAMA)
Response rate of SARS-CoV-2-specific neutralizing antibodies in serum samples | Measured through day 28
  Measured by neutralizing antibody assay (nAb)
Magnitude of SARS-CoV-2-specific antibody binding antibodies in serum samples | Measured through day 28
  Measured by binding antibody multiplex assay (BAMA)
Magnitude of SARS-CoV-2-specific neutralizing antibodies in serum samples | Measured through day 28
  Measured by neutralizing antibody assay (nAb)
Response rate of SARS-CoV-2-specific binding antibodies in nasal wash samples | Measured through day 28
  Measured by binding antibody multiplex assay (BAMA)
Magnitude of SARS-CoV-2-specific binding antibodies in nasal wash samples | Measured through day 28
  Measured by binding antibody multiplex assay (BAMA)
Frequency of leukocyte populations in peripheral blood | Measured through day 14
  Measured by flow cytometry
Transcriptional profiles of peripheral blood leukocytes | Measured through day 14
  Measured by gene expression analysis by RNA sequencing, real-time PCR, single-cell proteogenomic profiling
Concentration of serum cytokines and other soluble factors | Measured through day 28
  Measured by multiplexed protein detection assays and/or enzyme-linked immunosorbent assays (ELISA)
Response rate of SARS-CoV-2-specific CD4+ and CD8+ T cells | Measured through day 28
  Measured by flow cytometry
Magnitude of SARS-CoV-2-specific CD4+ and CD8+ T cells | Measured through day 28
  Measured by flow cytometry
Functional profiling, including intracellular cytokine staining, of SARS-CoV-2-specific CD4+ and CD8+ T cells | Measured through day 28
  Measured by flow cytometry

SECONDARY OUTCOMES:
Quantitation of viral RNA in nasal swabs | Measured through day 28
  Measured by extraction of nucleic acid for analysis of microorganism RNA or DNA by qPCR and/or amplicon- or metagenomics-sequencing methods and subsequent gene and taxa-level bioinformatics analyses

CONTACTS AND LOCATIONS:
Overall Officials: Will Hahn, Study Chair — Fred Hutch; Amy Ward, Study Chair — Cape Town - Khayelitsha
Locations (52):
- United States (15):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - University of Miami Infectious Disease Research Unit at Jackson Memorial Hospital CRS, Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - New Orleans Adolescent Trials Unit CRS, New Orleans, Louisiana
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Argentina (2):
  - Fundacion Huesped CRS, Buenos Aires
  - Hospital General de Agudos JM Ramos Mejía CRS, Buenos Aires
- Gaborone CRS, Gaborone, Botswana
- Brazil (2):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- Malawi CRS, Lilongwe, Malawi
- Merida CRS, Mérida, Mexico
- Peru (4):
  - CITBM - UNIDEC, Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales CRS, Bellavista
  - Asociacion Civil Selva Amazonica (ASCA) CRS, Iquitos
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
- South Africa (19):
  - Groote Schuur HIV CRS, Cape Town
  - Khayelitsha CRS / (CIDRI UCT), Cape Town
  - Masiphumelele Clinical Research Site (MASI) CRS, Cape Town
  - Chatsworth CRS, Chatsworth
  - Botha's Hill CRS, Durban
  - CAPRISA eThekwini CRS, Durban
  - Vulindlela CRS, Durban
  - Ndlovu Research Centre CoVPN CRS, Elandsdoorn
  - Isipingo CRS, Isipingo
  - Kliptown Soweto CRS, Johannesburg
  - Soweto HVTN CRS, Johannesburg
  - Aurum Institute Klerksdorp CRS, Klerksdorp
  - Qhakaza Mbokodo Research Clinic CRS, Ladysmith
  - MeCRU CRS, Medunsa
  - Nelson Mandela Academic Research Unit CRS, Mthatha
  - Rustenburg CRS, Rustenburg
  - Setshaba Research Centre CRS, Soshanguve
  - Tembisa Clinic 4 CoVPN CRS, Tembisa
  - Tongaat CRS, Tongaat
- National Institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC) Network CRS, Mbeya, Tanzania
- Zambia (3):
  - Matero Reference Clinic CRS, Lusaka
  - Zambia Emory HIV Research Project - Lusaka CoVPN CRS, Lusaka
  - Zambia Emory HIV Research Project - Ndola CoVPN CRS, Ndola
- Zimbabwe (3):
  - St Mary's CRS, Chitungwiza
  - Milton Park CRS, Harare
  - Seke South CRS, Harare